CLINICAL TRIAL: NCT00173537
Title: Genetic Research of Bone Morphogenetic Protein Receptor-II Gene in Taiwanese Patient With Primary Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 9461700712
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Pulmonary Hypertension
Keywords: idiopathic pulmonary artery hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Who Masked: Investigator

ARMS (1):
- other (Other)
  Interventions: Procedure: for BMPR II study; Genetic: BMPRII

INTERVENTIONS:
Procedure: for BMPR II study
Genetic: BMPRII

SUMMARY:
Primary pulmonary hypertension (PPH) is a rare lung disorder in which the blood pressure in the pulmonary artery rises far above normal levels for no apparent reason. The pulmonary artery is a blood vessel carrying oxygen-poor blood from the right ventricle (one of the heart's pumping chambers) to the lungs. In the lungs, the blood picks up oxygen, then flows to the heart's left side, where the left ventricle pumps it to the rest of the body through the aorta. In the United States, an estimated 500 to 1,000 new cases of primary pulmonary hypertension are diagnosed each year. The greatest number is reported in women between ages 20 and 40. However, men and women in all age ranges as well as very young children can develop PPH. Researchers have identified more than 40 BMPR2 mutations that can cause primary pulmonary hypertension. Many of these mutations introduce a stop signal that halts protein production prematurely, decreasing the amount of functional BMPR2 protein. Other mutations prevent the BMPR2 protein from reaching the cell surface, or alter its structure so it cannot form a complex with other proteins. It remains unclear how BMPR2 mutations cause primary pulmonary hypertension. Researchers suggest that a mutation in this gene prevents cell death or promotes cell proliferation, resulting in an overgrowth of cells in the blood vessels of the lungs. Cell overgrowth can narrow the diameter of the vessels, restricting blood flow and resulting in elevated blood pressure. However, it has not yet been reported regarding the genetic variants in Taiwan. Further details have been described in this project proposal.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as idiopathic pulmonary artery hypertension and associated family

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2005-07; Primary Completion 2009-11 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
all cause follow up | eight years
  all cause follow up

CONTACTS AND LOCATIONS:
Overall Officials: Hsao-Hsun Hsu, MD, Principal Investigator — Department of Surgery, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- See also: National Taiwan University Hospital Research Ethics Committee — http://www.ntuh.gov.tw/RECO/en/default.aspx